CLINICAL TRIAL: NCT02113826
Title: A Phase II Trial of Pazopanib in Patients With Metastatic Alveolar Soft Part Sarcoma
Brief Title: Pazopanib for Metastatic Alveolar Soft Part Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Asan Medical Center (Other); Samsung Medical Center (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Tae Min Kim, MD, PhD, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200240
Record Dates: First submitted 2014-04-09; First posted 2014-04-15 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Metastatic Alveolar Soft Part Sarcoma
Keywords: Pazopanib; Alveolar soft part sarcoma
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib (Experimental): Pazopanib 800mg po qd until disease progression
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib 800mg qd daily for 4 weeks = 1 cycle

SUMMARY:
Alveolar soft part sarcoma (ASPS), a rare subset of STS (<1%) harbors t(X;17)(p11;q25) translocation and produces resultant ASPL-TFE3 fusion protein. Due to its nature of high expression of angiogenic factors, sunitinib and cediranib produced overall response rates of 55% and 43%, respectively. However, the efficacy of pazopanib is unknown in metastatic ASPS.

DETAILED DESCRIPTION:
Pazopanib, a multi-targeted anti-angiogenesis inhibitor significantly prolonged progression-free survival (PFS) in patients with metastatic soft-tissue sarcoma (STS) after failure to anthracycline-based regimen (pazopanib vs placebo, 4.6 vs 1.6 months, HR=0.31, 95% CI 0.24-0.40; P < .0001). Regarding sunitinib (continuous daily dose of 37.5mg), after a median duration of 10 months, median OS and PFS were 19 months and 17 months, respectively in a small retrospective study (ASPS, N=9). With regard to cediranib, 6-month PFS was over 60%. In addition, randomized phase II trial of sunitinib vs cediranib with cross-over at disease progression was recently initiated (NCT01391962). However, the efficacy of pazopanib is unknown in metastatic ASPS.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of alveolar soft part sarcoma harboring TFE3 fusion at stage IV or at relapse
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Measurable lesion defined by RECIST v1.1
* Chemo-naïve or prior chemotherapies
* Adequate organ function

Exclusion Criteria:

* Prior malignancies
* Active CNS disease
* High-risk for gastrointestinal bleeding
* Significant cardiovascular disease
* Uncontrolled hypertension
* Bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-04; Primary Completion 2016-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | One year
  ORR based on RECIST v1.1

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | One year
  Safety based on CTCAE v4.0
Progression-free survival | 6 month
Overall survival | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim M, Kim TM, Keam B, Kim YJ, Paeng JC, Moon KC, Kim DW, Heo DS. A Phase II Trial of Pazopanib in Patients with Metastatic Alveolar Soft Part Sarcoma. Oncologist. 2019 Jan;24(1):20-e29. doi: 10.1634/theoncologist.2018-0464. Epub 2018 Sep 25. PMID 30254189